CLINICAL TRIAL: NCT06762405
Title: PRODIGE 90 - (FFCD 2204) - PREDIR-NEOREC Neoadjuvant Dostarlimab with Short Course Radiotherapy in a Watch-and-wait Strategy for Microsatellite Unstable or Mismatch Repair-deficient Locally Advanced Rectal Cancer Patients: a Randomized Phase II Trial Phase II Randomized Study Non-comparative - Multicenter
Brief Title: PRODIGE 90 - (FFCD 2204) Neoadjuvant Dostarlimab with Short Course Radiotherapy in a Watch-and-wait Strategy for Microsatellite Unstable or Mismatch Repair-deficient Locally Advanced Rectal Cancer Patients
Acronym: PREDIR-NEOREC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DROUILLARD PHRCK 2023-1
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Rectal Adenocarcinoma with Mismatch-repair Deficient (dMMR)/ Microsatellite Instability-high (MSI-H)
MeSH Terms: interventions — Radiotherapy; dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiotherapy followed by Dostarlimab arm (Experimental)
  Interventions: Radiation: radiotherapy; Drug: Dostarlimab; Biological: Biological study on circulating tumor DNA (optional for the patient)
- Dostarlimab alone arm (Active Comparator)
  Interventions: Drug: Dostarlimab; Biological: Biological study on circulating tumor DNA (optional for the patient)

INTERVENTIONS:
Radiation: radiotherapy — short course of radiotherapy (5 grays × 5 days)
  Arms: Radiotherapy followed by Dostarlimab arm
Drug: Dostarlimab — dostarlimab 500 mg intravenous infusion every 3 weeks for 6 months (nine cycles)
Biological: Biological study on circulating tumor DNA (optional for the patient) — * Tissue collection (3 time points: baseline, w12 and 25) for:
  * Exome (on tumor and normal tissue),
  * 3'RNAseq,
  * Hiplex Immunofluorescence
  * In addition, 48 patients will be tested for Spatial transcriptomics assuming that 24 patients may have non-complete response and/or local recurrence and/or metastatic recurrence and will be paired with 24 patients with complete response and free of any disease at 2 years.
  * Blood collection (5 time points: baseline, w3, 6, 12 and 24) for:
  * ctDNA
  * Cytokine dosage
  * Proteomic analyses
  * Stool collection (3 time points: baseline, w3 and 24) for:
  Microbiota analyses

SUMMARY:
Total neoadjuvant treatment (TNT) including radiotherapy and induction or consolidation systemic chemotherapy has become the standard treatment for patients with stage II and III rectal adenocarcinoma. Along with the improvement of DFS, this preoperative treatment has paved the way to a paradigm-shifting nonoperative management. Indeed, rectal preservation has become a new goal for patients without detectable residual cancer after TNT with the option to reserve surgery for those with cancer regrowth (25-40%). Five to 10% of non-metastatic rectal cancer patients are molecularly characterized as microsatellite unstable (MSI) or mismatch repair-deficient (dMMR), and present a decreased response to systemic chemotherapy. As this tumor phenotype is associated with high immunogenicity, immunotherapy with anti-PD1 molecules has recently emerged as the new standard first line treatment in the metastatic setting, with long duration of cancer control for at least 40% of patients. In patients with localized rectal tumors, it has been suggested that immunotherapy alone may induce complete clinical response and may allow these patients to be considered for nonoperative therapeutic approaches.

Finally, given the efficacy of immunotherapy in MSI rectal patients, we did not want to differ for 5 weeks this treatment with the risk of disease progression by given long-course RT. In the present trial, radiotherapy is evaluated as a " potentiating " treatment for immunotherapy rather than as a " local treatment " in a TNT strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically proven rectal adenocarcinoma with Mismatch-repair Deficient (dMMR)/ microsatellite instability-high (MSI-H). Tumour status (dMMR/MSI-H) should be determined using both IHC (Immunohistochemistry) and PCR (polymerase chain reaction) or NGS (Next-Generation sequencing)
* Stage II or III and middle and lower third rectal adenocarcinoma (diagnosed on the basis of standard clinical and MRI criteria)
* WHO performance status 0 or 1
* Adequate liver function: AST and ALT ≤ 5 x ULN (upper normal limit), total bilirubin ≤ 35 μM/L, albumin ≥ 28 g/L and Child-Pugh A score (if cirrhosis associated)
* Adequate hematological and renal function (hemoglobin > 9 g/dl, platelets > 100 G/L, ANC ≥ 1.5 G/L) and renal function (creatinine clearance ≥ 40ml/min according to MDRD formula)
* Women of childbearing potential must agree to use contraception during the trial treatment and for at least 4 months after discontinuation of the experimental treatments. Men who have sex with women of childbearing potential must agree to use contraception during treatment and for at least 4 months after discontinuation of the experimental treatments
* Ability of patient to understand, sign and date the informed consent form before any study specific screening procedures
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Stage IV and upper third rectal adenocarcinoma (above 10 cm from the anal verge or sus-peritoneal on standard clinical and MRI criteria)
* Patients who have already received immunotherapy, chemotherapy or radiotherapy for rectal cancer
* Persistent toxicities related to prior treatment of grade greater than 1
* Participant has an active infection requiring systemic therapy within 1 week prior to the anticipated first dose of study treatment
* Contraindication to pelvic radiotherapy
* Hypersensitivity to dostarlimab or any of its excipients
* Allergy to any component of Chinese hamster ovary cells
* History of severe active life-threatening autoimmune disease
* History of uncontrolled or symptomatic cardiac disease.
* Interstitial lung disease
* Uncontrolled central nervous system metastases or carcinomatous meningitis
* Patient has documented presence of HBsAg [or HBcAb] at screening or within 3 months prior to first dose of study intervention
* Patient has a positive HCV antibody test result at screening or within 3 months prior to first dose of study intervention. NOTE: Participants with a positive HCV antibody test result due to prior resolved disease can be enrolled, only if a confirmatory negative HCV RNA test is obtained
* Patient has a positive HCV RNA test result at Screening or within 3 months prior to first dose of study intervention. NOTE: The HCV RNA test is optional and participants with negative HCV antibody test are not required to undergo HCV RNA testing as well
* Known HIV infection
* Vaccinations (live vaccine) within 14 days prior to start of treatment
* Immunosuppression, including subjects with conditions requiring systemic corticosteroid treatment (>10 mg/day prednisone equivalent)
* Active autoimmune disease requiring systemic treatment (vitiligo excluded) in the past 2 years or recent receipt within the previous 7 days of immunosuppressive therapy
* History of organ transplantation
* Pregnant or breastfeeding women
* Patient has experienced any of the following with prior immunotherapy: any immune-related AE (irAE) of Grade 3 or higher, immune-related severe neurologic events of any grade (e.g., myasthenic syndrome/myasthenia gravis, encephalitis, Guillain-Barré Syndrome, or transverse myelitis), exfoliative dermatitis of any grade (Stevens-Johnson Syndrome, toxic epidermal necrolysis, or drug reaction with eosinophilia and systemic symptoms [DRESS] syndrome), or myocarditis of any grade. Non-clinically significant laboratory abnormalities are not exclusionary
* Any progressive disease that has not been balanced over the last 6 months: hepatic insufficiency, renal insufficiency, respiratory insufficiency, etc
* Other cancer treated within the last 5 years except in situ cervical carcinoma or basocellular/ spinocellular carcinoma or a cancer of the lynch syndrome spectrum considered cured at the time of inclusion
* Major surgery within 4 weeks before inclusion
* Persons deprived of liberty or under guardianship or incapable of giving consent
* Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol or follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Treatment strategy failure (TSF) rate. | at 24 months
  TSF is defined as the rate of patients without a clinical complete response (cCR) regarding all the clinical exams (Digital Rectal Exam, MRI and Endoscopy) and those with a cCR but with local or metastatic recurrence or local regrowth within 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France